CLINICAL TRIAL: NCT00425763
Title: Efficacy of Amodiaquine-artesunate in the Treatment of Symptomatic, Uncomplicated Plasmodium Falciparum Malaria Among 6-59 Month Old Children at an IPTi Site in Rural Western Kenya
Brief Title: Efficacy of Amodiaquine-artesunate in Children Aged 6-59 Months With Uncomplicated P. Falciparum Malaria
Acronym: IPTi DRWG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-5022; KEMRI-SSC-1190
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Malaria
Keywords: malaria; efficacy; intermittent preventive therapy in infants; drug resistance
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AQAS (Experimental)
  Interventions: Drug: AQAS

INTERVENTIONS:
Drug: AQAS — AQAS dosed by body weight, on days 0, 1, 2

SUMMARY:
We will be studying the clinical efficacy of amodiaquine-artesunate currently being studied in an intermittent preventive therapy in infants (IPTi)trial in the same area in order to correlate preventive efficacy seen in IPTi with efficacy for treatment of symptomatic malaria for each regimen.

DETAILED DESCRIPTION:
We propose to conduct an amodiaquine-artesunate efficacy trial at Bondo District Hospital in Kenya. The results will enable us to better interpret the results of the main IPTi trial. We will assess the efficacy of a three day course of amodiaquine plus three days of artesunate (AQ3/AS3) for the treatment of symptomatic, uncomplicated P. falciparum infections. Study subjects are febrile children, 6-59 months old, with laboratory-confirmed uncomplicated P. falciparum infections. Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy. Children will be followed closely for signs of drug failure or recrudescence, and any children failing therapy will be treated with Coartem or, if severe, with quinine. We will also perform drug resistance testing on parasite samples from children with treatment failure. The results of this efficacy trial will allow us to assist policymakers in deciding what drugs should be used for IPTi, should it be adopted into national policy.

ELIGIBILITY:
Inclusion Criteria:

* age 6-59 months
* axillary temperature ≥ 37.5º C, or history of fever in previous 24 hours
* weight ≥ 5.0 kg
* slide-confirmed infection with P. falciparum
* parasitemia 2000-200,000 asexual forms per μl
* ability and willingness to attend stipulated follow-up visits

Exclusion Criteria:

* signs or symptoms of severe disease
* weight-for-age ≤ 3rd percentile on Kenya growth charts
* slide confirmed infection with any other Plasmodium spp., besides falciparum
* severe anemia, defined as Hb < 7 g/dl
* known hypersensitivity to any of the drugs being tested
* enrolled in IPTi trial
* known chronic disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
28 Day Adequate Clinical and Parasitological Response, Early Treatment Failure, Late Clinical Failure, Late Parasitological

SECONDARY OUTCOMES:
Side effects
Molecular markers of drug resistance

CONTACTS AND LOCATIONS:
Overall Officials: Meghna Desai, PhD, Principal Investigator — Centers for Disease Control and Prevention; Mary Hamel, MD, Principal Investigator — Centers for Disease Control and Prevention; Patrick Kachur, MD, MPH, Study Chair — Centers for Disease Control and Prevention; Robert Newman, MD, MPH, Study Chair — Centers for Disease Control and Prevention; Larry Slutsker, MD, MPH, Study Chair — Centers for Disease Control and Prevention; Julie Thwing, MD, Study Director — Centers for Disease Control and Prevention; Christopher O Odero, Study Director — CDC/KEMRI
Locations (1):
- Bondo District Hospital, Kisumu, Kenya